CLINICAL TRIAL: NCT05807048
Title: A Single-Arm Phase 2 Study of Daratumumab Subcutaneous (SC) in Previously Treated STK11/LKB1 Mutated Non-small Cell Lung Cancer
Brief Title: Daratumumab in STK11 Mutated NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-01512
Record Dates: First submitted 2023-03-29; First posted 2023-04-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer With STK11/LKB1 Mutation
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with STK11/LKB1-Mutated NSCLC (Experimental): Participants will receive daratumumab 1800mg and hyaluronidase 30,000 units (combined product DARZALEX Faspro) administered subcutaneously per the following dosing schedule:
  * Once per week for 8 administrations (Week 1-8)
  * Once every two weeks for 8 administrations (Week 9-16)
  * Once every 4 weeks until disease progression or unacceptable toxicity.
  Interventions: Drug: Daratumumab and Hyaluronidase-fihj; Drug: Pre-Intervention Medication; Drug: Post-Intervention Medication

INTERVENTIONS:
Drug: Daratumumab and Hyaluronidase-fihj — DARZALEX FASPRO (daratumumab and hyaluronidase-fihj) injection for subcutaneous use. Supplied as individually packaged single-dose vials providing 1,800 mg of daratumumab and 30,000 units of hyaluronidase per 15 mL.
  Other Names: DARZALEX FASPRO
Drug: Pre-Intervention Medication — The following pre-medications will be administered 1-3 hours before each dose of DARZALEX FASPRO:
  * Acetaminophen 650 to 1,000 mg orally
  * Diphenhydramine 25 to 50 mg (or equivalent) orally or intravenously
  * Montelukast 10mg PO prior to DARZALEX FASPRO®.
  * Methylprednisolone 100 mg (or equivalent) orally or intravenously
Drug: Post-Intervention Medication — The following post-medications will be administered:
  * Methylprednisolone 20 mg (or an equivalent dose of an intermediate- or long acting corticosteroid) orally for 2 days starting the day after the administration of DARZALEX FASPRO®.
  * Patients with a history of chronic obstructive pulmonary disease will be prescribed short and long-acting bronchodilators and inhaled corticosteroids.
  * Antiviral prophylaxis for herpes zoster reactivation must be initiated within one week of daratumumab hyaluronidase-fihj administration and continued for 3 months following the end of treatment.

SUMMARY:
This is a single-arm study of daratumumab in metastatic non-small cell lung cancer (NSCLC) patients with an STK11/LKB1 mutation. Patients will have received previous standard of care treatment including chemotherapy, immunotherapy and targeted therapy. Patients will be treated with the standard subcutaneous dosing of daratumumab (weekly for 8 administrations, then every 2 weeks for 8 administrations then every 4 weeks until progression). All follow-up visits and imaging will be performed as per standard of care. This is a signal finding study and an overall response rate ≥20% is considered clinically meaningful.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age and satisfy the legal age of consent in the jurisdiction in which the study is being conducted.
* Participant must have histologically or cytologically confirmed NSCLC that is metastatic or unresectable.
* Participants must have either progressed after prior immunotherapy with a PD-(L)1 inhibitor, platinum doublet chemotherapy and standard of care targeted therapy (if presence of an activating mutation is identified) for metastatic disease, be ineligible for, or have refused all therapeutic options. In cases where participants refuse currently available therapeutic options, this must be documented in the study records.
* Participants must have previously identified STK11/LKB1 mutation (identified locally in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory [or equivalent])
* Participant must have organ and bone marrow function as follows:

  * Hemoglobin ≥9 g/dL
  * Absolute blood neutrophil count (ANC) ≥1.5 x 109 /L
  * Platelets ≥75 x 109 /L
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 x upper limit of normal (ULN)
  * Total bilirubin =1.5 x ULN; participants with Gilbert's syndrome can enroll if conjugated bilirubin is within normal limits.
  * Serum creatinine <1.5 x ULN or if available, calculated or measured creatinine clearance; >50 mL/min/1.73 m2
* Before enrollment, a woman must be either:

  * Not of childbearing potential: postmenopausal (>45 years of age with amenorrhea for at least 12 months); permanently sterilized (eg, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy,
  * Of childbearing potential and practicing a highly effective method(s) of birth control consistent with local regulations regarding the use of birth control methods for participants participating in clinical studies, described as follows: practicing true abstinence (when this is in line with the preferred and usual lifestyle of the participant), which is defined as refraining from heterosexual intercourse during the entire period of the study, including up to 6 months after the last dose of study drug is given; OR have a sole partner who is vasectomized; OR practicing 2 methods of contraception, including one highly effective method (ie, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device [IUD] or intrauterine system [IUS]), AND, a second method, (eg, condom with spermicidal foam/gel/film/cream/suppository or occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository).
  * Note: If the childbearing potential changes after start of the study (eg, woman who is not heterosexually active becomes active, postmenopausal woman experiences menarche) the woman must begin a highly effective method of birth control, as described above.
* A woman of childbearing potential must have a negative serum (β-human chorionic gonadotropin [β-hCG]) at Screening and a negative urine or serum pregnancy test within 24 hours before the first dose of study drug.
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study drug.
* A man who is sexually active with a woman of childbearing potential must agree to use a condom and his partner must also be practicing a highly effective method of contraception (ie.. established use of oral, injected or implanted hormonal methods of contraception; placement of an IUD or IUS). If the participant is vasectomized, he must still use a condom, but his female partner is not required to use contraception. The participant must also not donate sperm during the study and for 6 months after receiving the last dose of study drug.
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, including the agreement by both male and female participants to continue contraception throughout the study and through 6 months after the last dose of study drug.
* Each participant must sign an informed consent form (ICF) indicating that he or she understands the study's purpose and the procedures required for the study and is willing to participate in the study, including the requirement to provide information during the Follow-up period.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Participant has uncontrolled inter-current illness, including but not limited to poorly controlled hypertension or diabetes, ongoing or active systemic infection (ie, has discontinued all antibiotics for at least one week prior to first dose of study drug), diagnosed or suspected viral infection (except for HIV), or psychiatric illness/social situation that would limit compliance with study requirements, including ability to self-care for anticipated toxicities (eg. rash or paronychia).
* Participants with medical conditions requiring chronic continuous oxygen therapy are excluded.
* Participants with a history of chronic obstructive pulmonary disease (COPD) with grade ≥3 breathlessness on the modified medical research council (mMRC) dyspnea scale are excluded.
* Have known moderate or severe persistent asthma within the past 2 years, or current uncontrolled asthma of any classification.
* Participant has a history of clinically significant cardiovascular disease including, but not limited to:

  * Diagnosis of deep vein thrombosis or pulmonary embolism within 4 weeks prior to the first dose of study drug, or any of the following within 6 months prior to the first dose of study drug: myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary/peripheral artery bypass graft, or any acute coronary syndrome. Clinically non-significant thrombosis, such as non-obstructive catheter-associated clots, are not exclusionary.
  * Prolonged QTcF interval >480 msec or clinically significant cardiac arrhythmia or electrophysiologic disease (eg, placement of implantable cardioverter defibrillator or atrial fibrillation with uncontrolled rate). Note: Participants with cardiac pacemakers who are clinically stable are eligible.
  * Uncontrolled (persistent) hypertension: systolic blood pressure >180 mm Hg; diastolic blood pressure >100 mm Hg
  * Congestive heart failure defined as New York Heart Association (NYHA) class III-IV or Hospitalization for congestive heart failure (any NYHA class) within 6 months of study Day 1
  * Pericarditis/clinically significant pericardial effusion
  * Myocarditis
* Participant has had prior chemotherapy, targeted cancer therapy, or treatment with an investigational anti-cancer agent within 2 weeks or 4 half-lives, whichever is longer, before the first administration of study drug; or participant has received prior immunotherapy within 6 weeks before the first administration of study drug. For agents with long half-lives, the maximum required time since last dose is 4 weeks. Toxicities from previous anticancer therapies should have resolved to baseline levels or to Grade 1 or less, (except for alopecia [any grade], Grade ≤2 peripheral neuropathy, and Grade <2 hypothyroidism stable on hormone replacement). Autoimmune toxicities from previous immunotherapy must be fully resolved to baseline levels.
* Localized, radiotherapy for palliative purposes must be completed at least 7 days prior to treatment with daratumumab and hyaluronidase.
* Participants with untreated brain metastases. Participants with locally treated metastases that are clinically stable and asymptomatic for at least 2 weeks and who are off or receiving low-dose corticosteroid treatment (≤10 mg prednisone or equivalent) for at least 2 weeks prior to study treatment are eligible.
* Participant has leptomeningeal disease.
* Participant has an active malignancy other than the disease under study requiring treatment or a history of malignancy unless all treatment of that malignancy was completed at least 2 years before consent and the patient has no evidence of disease before the date of randomization. Exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator is considered cured with minimal risk of recurrence within 3 years.
* Participant has known allergies, hypersensitivity, or intolerance to daratumumab or hyaluronidase or its excipients.
* Participants with known allergies, hypersensitivity to any component of montelukast.
* Participant has received an investigational drug (including investigational vaccines but not including anti-cancer therapy [refer to Exclusion Criterion #3]) or used an invasive investigational medical device within 6 weeks before the planned first dose of study drug.
* Participant is a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of study drug.
* Participant has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
* Participant has at Screening:

  * Positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg) Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
  * Positive hepatitis C antibody (anti-HCV). Note: Participants with a prior history of HCV, who have completed antiviral treatment and have a sustained virologic response, defined as aviremia at least 12 weeks after completion of antiviral therapy are eligible. Patients who completed treatment for hepatitis C at least 6 months prior to screening and have no detectable circulating HCV during screening may participate in the study. Such patients will be required to undergo regular assessments for HCV reactivation during the study and are to be withdrawn from the study if he/she test positive at any time during the study.
  * Other clinically active infectious liver disease.
* Seropositive for human immunodeficiency virus.
* Participant has had prior therapy with daratumumab.
* Have had major surgery within 2 weeks before randomization or will not have fully recovered from surgery, or has surgery planned during the time the patient is expected to participate in the study or within 2 weeks after the last dose of study treatment. Note, patients with planned surgical procedures to be conducted under local anesthesia may participate.
* Have received vaccination with live attenuated vaccines within 4 weeks of first study agent administration.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) based on RECIST 1.1 Criteria | Up to Month 24
  ORR is the percentage of patients who best response recorded from study enrollment until disease progression is a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, where:
  CR = disappearance of all target lesions; and PR = at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Number of Adverse Events | Up to Month 24
  Number of adverse events as defined by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Number of Severe Adverse Events | Up to Month 24
  Number of grade 3-5 adverse events as defined by NCI-CTCAE version 5.0.
Number of Adverse Events Attributed to Study Drugs | Up to Month 24
  Number adverse events related to study drugs as defined by NCI-CTCAE version 5.0.
Percent of Participants who Experience Complete Response (CR) | Up to Month 24
  Percent of participants who experience CR according to RECIST 1.1, where CR = disappearance of all target lesions.
Percent of Participants who Experience Partial Response (CR) | Up to Month 24
  Percent of participants who experience PR according to RECIST 1.1, where PR = at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Percent of Participants who Experience Stable Disease (SD) | Up to Month 24
  Percent of participants who experience SD according to RECIST 1.1, where SD = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as reference the smallest sum diameters while on study.
Duration of Response (DoR) | Up to Month 24
  DoR is the time from randomization to disease progression or death in patients who achieve CR or PR according to RECIST 1.1.
Progression-Free Survival (PFS) | Up to Month 24
  PFS is the duration of the date of first treatment to the date of first documented evidence of progressive disease or death, whichever comes first.
Overall Survival (OS) | Up to Month 24
  OS is the duration of the date of first treatment to the date of the participant's death.

CONTACTS AND LOCATIONS:
Overall Officials: Salman Punekar, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: sally.lau@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted upon reasonable request. Requests should be directed to sally.lau@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.